CLINICAL TRIAL: NCT01960881
Title: Canadian Real Life Evaluation of the Effect of Diet and Exercise in Prostate Cancer Patients Managed With Lupron (CRONOS II)
Brief Title: Evaluation of Diet and Exercise in Prostate Cancer Patients
Acronym: CRONOS II
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Collaborators: JSS Medical Research; CMX Research Inc.; Canadian Urology Research Consortium (Unknown)
Responsible Party: Sponsor
Other Study IDs: P14-096
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prostate Cancer Patients: Prostate Cancer Patients

SUMMARY:
Canadian Real Life Evaluation of the Effect of Diet and Exercise in Prostate Cancer Patients Managed with Lupron.

DETAILED DESCRIPTION:
This is a study utilizing a prospective cohort design. Patients with Prostrate cancer (PCa) who are prescribed Lupron will be entered into the study cohort and will be followed for a maximum of 18 months with recommended assessments at 3, 6, 12 and 18 months after Day 1. Treatment of the patients and follow up will be according to the physicians' judgment, regional regulations and the product monograph.

ELIGIBILITY:
Inclusion Criteria:

i. Adult ≥ 18 years old

ii. Has provided written informed consent allowing the use of their data for the study and providing permission for contact by the study personnel.

iii. Diagnosed with PCa.

iv. Prescribed Lupron as part of his treatment by his treating physician.

Exclusion Criteria:

i. Patient cannot or will not sign informed consent.

ii. Presence of other condition that, in the opinion of the treating physician, prohibits the patient from participating in the study or obscures the assessment of the treatment of PCa.

iii. More than 6 months of therapy if currently on continuous Luteinizing hormone-releasing hormone (LHRH) treatment.

iv. If at study enrollment the intent is to only prescribe 1 dose of Lupron (leuprolide acetate)

Ages: 18 Years to 99 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled from the offices of University or community urologists/radio-oncologists across Canada treating patients with PCa
Sampling Method: Non-Probability Sample
Enrollment: 1331 (Actual)
Dates: Start 2013-09-19 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Changes in the patient quality of life (QoL) using the Medical Outcomes Study Short Form - 36 (SF-36) | From Month 0 to Month 18
  The SF-36 Health is a 36-item general health self-administered questionnaire consisting of 8 scales measuring Physical Function, Physical Role limitations, Vitality, General Health, Pain, Social Function, Emotional Role limitations, and Mental Health.
Change in exercise duration | From Month 0 to Month 18
  Assessed at every visit what was the amount of various types of exercise performed in the previous month.
Change in dietary habits | From Month 0 to Month 18
  Assessed at every visit to what extent patient's complied with the Canadian Food Guide's recommendation for each of the four food group servings in the previous week.

SECONDARY OUTCOMES:
Change in the patient quality of life (QoL) using the Medical Outcomes Study Short Form - 36 (SF-36) | From Month 0 to follow-up visits 3,6 and 12 months
  The SF-36 Health is a 36-item general health self-administered questionnaire consisting of 8 scales measuring Physical Function, Physical Role limitations, Vitality, General Health, Pain, Social Function, Emotional Role limitations, and Mental Health.
Change in weight | From Month 0 to Month 18
  Change from Baseline is calculated as the post-Baseline value minus the Baseline value.
Change in Body Mass Index (BMI) | From Month 0 to Month 18
  BMI is a measure of body fat based on weight in relation to height. Change from Baseline is calculated as the post-Baseline value minus the Baseline value.
Changes in the University of California Los Angeles Prostate Cancer Index (UCLA-PI) | From Month 0 to Month 18
  A validated questionnaire designed to measure quality of life in patients with prostate cancer. It consists of 20 questions that assess urinary, sexual, bowel and hormonal function and impairment in patients with prostate cancer.
Changes in the sexual function using the International Index of Erectile Function (IIEF-5) | From Month 0 to Month 18
  An abridged 5 item self-administered questionnaire assessing the presence and severity of erectile dysfunction (for patients enrolled prior to protocol amendment 2)
Number of patients with Adverse Events | From Month 0 to Month 18
  Adverse events which lead to discontinuation of prescribed treatment under observation, will be coded according to the Medical Dictionary for Regulatory Activities (MeDRA) dictionary of terms
Changes in the patient's medical condition | From Month 0 to Month 18
  Any change in the patient's medical condition including new onset or worsening of medical conditions.
Proportion of patients with castrate levels of testosterone and undetectable levels of Prostatic Specific Antigen (PSA) at 18 months of treatments. | From Month 0 to Month 18
  The PSA test measures the level of PSA in a man's blood. For this test, a blood sample is sent to a laboratory for analysis. The results are usually reported as nanograms of PSA per milliliter (ng/mL) of blood. A testosterone test checks the level of this male hormone (androgen) in the blood.
Leuprolide Acetate Utilization | From Month 0 to Month 18
  Utilization of Leuprolide Acetate will be assessed.
Changes in the Doctor-Patient communication (for patients enrolled prior to protocol amendment 2) | From Month 0 to Month 18
  This will be ascertained with the Doctor-Patient Communication/Doctor's Questionnaire and the Doctor-Patient Communication/Patient's Questionnaire that are validated questionnaires developed by the College of Physicians of Quebec
Caregiver Quality of Life (for patients enrolled under protocol amendment 1) | From Month 0 to Month 18
  Measured with the Caregiver Quality of Life Index - Cancer scale (CQOLC). This is a 35 item questionnaire that measures the quality of life of individuals caring for cancer patients.
Assessment of Financial Burden on Patient's Family (for patients enrolled under protocol amendment 1) | Up to Month 18
  Measured with a self-reported questionnaire.
Lupron Cares Patient Support Program | Up to Month 18
  Enrollment and use will be assessed for the patient support program.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (50):
- Canada (50):
  - Exdeo Clinical Research Inc /ID# 116040, Abbotsford, British Columbia
  - Southern Interior Medical Research /ID# 116025, Kelowna, British Columbia
  - Dr. J. Paul Whelan, Inc. /ID# 120415, Victoria, British Columbia
  - CancerCare Manitoba /ID# 135976, Winnipeg, Manitoba
  - Saint John Regional Hospital /ID# 141302, Saint John, New Brunswick
  - QE II Health Sciences Centre /ID# 118941, Halifax, Nova Scotia
  - The Male/Female Hlth and Res /ID# 116042, Barrie, Ontario
  - The Male/Female Hlth and Res /ID# 124295, Barrie, Ontario
  - Edward F.A. Woods Medicine Professional Corporation /ID# 120695, Belleville, Ontario
  - Jonathan Giddens Medicine /ID# 116023, Brampton, Ontario
  - Brantford Urology Research /ID# 116026, Brantford, Ontario
  - G. Kenneth Jansz Medicine Professional Corporation /ID# 116024, Burlington, Ontario
  - William R. Love, Medicine, Professional Corporation /ID# 116035, Burlington, Ontario
  - Northern Urology Centre /ID# 141391, Greater Sudbury, Ontario
  - St. Joseph's Healthcare /ID# 163973, Hamilton, Ontario
  - Queen's University /ID# 137983, Kingston, Ontario
  - London Health Sciences Center /ID# 118940, London, Ontario
  - DiCostanzo, Markham, CA /ID# 137272, Markham, Ontario
  - Mor Urology Inc /ID# 116027, Newmarket, Ontario
  - Stanley Flax Medical Prof Corp /ID# 116022, North YORK, Ontario
  - Fe/Male Health Centers /ID# 116020, Oakville, Ontario
  - The Ottawa Hospital /ID# 132329, Ottawa, Ontario
  - Dr. Sean Pierre Medicine Professional Corporation /ID# 137986, Ottawa, Ontario
  - Kawarth Urology Associates /ID# 116041, Peterborough, Ontario
  - The Medical Centre /ID# 128278, Peterborough, Ontario
  - Abara Medicine Professional Corporation /ID# 137270, Richmond Hill, Ontario
  - Dr. Petar Erdeljan Medicine Professional Corporation /ID# 139641, Scarborough Village, Ontario
  - 1837206 Ontario Inc. /Id# 116038, Scarborough Village, Ontario
  - Urology and Male Fertility /ID# 116043, Scarborough Village, Ontario
  - Duplicate_Sunnybrook Health Sciences Ctr /ID# 136597, Toronto, Ontario
  - Princess Margaret Cancer Centre /ID# 137984, Toronto, Ontario
  - Toronto Urology Clin Study Grp /ID# 116044, Toronto, Ontario
  - Toronto West Urology Associates /ID# 116021, Toronto, Ontario
  - Toronto West Urology Associates /ID# 134134, Toronto, Ontario
  - Clinique d'urologie /ID# 116019, Chicoutimi, Quebec
  - CISSS - Hôpital de Gatineau /ID# 131309, Gatineau, Quebec
  - CISSS de la Monteregie /ID# 116036, Greenfield Park, Quebec
  - CISSS de la Monteregie /ID# 124296, Greenfield Park, Quebec
  - CISSS de la Monteregie /ID# 134137, Greenfield Park, Quebec
  - Clinique d'Urologie á Polyclinique Médicale Concorde /ID# 116037, Laval, Quebec
  - Hopital Cite-de-la-Sante /ID# 130951, Laval, Quebec
  - CHUM - Notre-Dame Hospital /ID# 137271, Montreal, Quebec
  - Montreal General Hospital - McGill University Health Center /ID# 141503, Montreal, Quebec
  - Jewish General Hospital /ID# 120416, Montreal, Quebec
  - Ultra-Med Research /ID# 116355, Pointe-Claire, Quebec
  - CHUS - Hopital Fleurimont /ID# 124275, Sherbrooke, Quebec
  - Ctr Sante et Services Sociaux /ID# 131230, Trois-Rivières, Quebec
  - Groupe De Recherche En Urologie De La Mauricie /ID# 116356, Trois-Rivières, Quebec
  - Clinique des Spécialités Chirurgicales de Val-d'Or /ID# 116039, Val-d'Or, Quebec
  - 9120-1947 Quebec Inc. /ID# 129151, Westmount, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P14-096&Latitude=&Longitude=&LocationName=#additional-resources-section